CLINICAL TRIAL: NCT06728475
Title: Effect Of Virtual Reality With Mirror Therapy on Upper Limb Functions in Children With Hemiplegic Cerebral Palsy
Brief Title: Virtual Reality With Mirror Therapy on Upper Limb Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Khalid Esmail Mohamed Mohamed, Effect Of Virtual Reality with Mirror Therapy on Upper Limb Functions in Children with Hemiplegic Cerebral Palsy, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KFSIRB200-254
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hemiplagia; Upper limb function; Virtual reality; Mirror therapy; Xbox 360
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) virtual reality group (Active Comparator): this group will receive virtual reality intervention plus designed physical therapy program
  Interventions: Device: virtual reality
- Group (B) mirror therapy group (Active Comparator): this group will receive mirror therapy intervention plus designed physical therapy program
  Interventions: Other: mirror therapy
- Group (C) the compound effect of virtual reality and mirror therapy group (Active Comparator): this group will receive virtual reality intervention , mirror therapy intervention plus designed physical threrapy program
  Interventions: Other: virtual reality with mirror therapy

INTERVENTIONS:
Device: virtual reality — In Xbox, we will choose suitable games that aim to improve upper limb function like boxing, Darts, tennis, goalkeeping, basketball, disc throwing, balling, and volleyball.
  The Kinect sensor has the advantage of auto adjustment of its camera according to the child's position and height that's to say the child can perform the game in sitting or standing according to their abilities.
  They will receive 30 minutes of VR intervention in addition to the time required for the designed physical therapy program.
  Arms: Group (A) virtual reality group
Other: mirror therapy — Mirror Therapy A mirror of 30 × 20 inches was used for the MT, which was large enough to cover the entire affected limb while still allowing the reflection of the non-affected limb to be seen. The child was seated in a chair with the forearms resting on the table. In the mid-sagittal plane, the mirror box was positioned at an angle of 70° to 80° to the trunk. The affected limb was placed behind the mirror. The child was asked to perform the exercises bilaterally and symmetrically as much as possible. Even if the affected side did not move easily or fully, the child was advised to synchronize the motions with both hands and arms. The researcher constantly reminded the child to concentrate on the movement of the non-affected limb in front of the mirror, which helped to increase the mirror illusion
  Arms: Group (B) mirror therapy group
Other: virtual reality with mirror therapy — group C will receive combined effect of both techniques (virtual reality and mirror therapy)
  Arms: Group (C) the compound effect of virtual reality and mirror therapy group

SUMMARY:
The goal of this clinical trial is to address the effect of (Virtual Reality) and (Mirror Therapy) together on upper limb function in hemiplegic Cerebral Palsy children , male or female ranged between 3 to 10 years of age

. The main question of the study is Are there any significant differences between the effects of virtual reality , mirror therapy and the combined effect of both techniques and on upper limb function in hemiplegic CP children?

Participants will be subdevided into three groups A , B ,C Group (A): will receive VR in addition to designed physical therapy program Group (B): will receive MT in addition to designed physical therapy program Group (C): will receive the compound effect of both techniques in addition to designed physical therapy program

DETAILED DESCRIPTION:
The goal of this clinical trial is to address the effect of (Virtual Reality) and (Mirror Therapy) together on upper limb function in hemiplegic Cerebral Palsy children , male or female ranged between 3 to 10 years of age

. The main question of the study is Are there any significant differences between the effects of virtual reality (VR), mirror therapy (MR) and the combined effect of both techniques (VR) and (MR) on upper limb function in hemiplegic CP children?

Participants will be subdevided into three groups A , B ,C Group (A): will receive VR in addition to designed physical therapy program Group (B): will receive MT in addition to designed physical therapy program Group (C): will receive the compound effect of both techniques in addition to designed physical therapy program

ELIGIBILITY:
Inclusion Criteria:

* Children will be included in the study if they fulfil the following criteria:

  1. A medical diagnosis of spastic hemiplegic CP made by pediatric neurologists.
  2. Children with spasticity grades ranged from 1 to 1+ according to MAS.
  3. Their age range from 4 to 10 years.
  4. Children level 1 and level 2 in gross motor functional classification (GMFC 1&2)

Exclusion Criteria:

* Children will be excluded from the study if:

  1. They had a permanent deformity (bony or soft tissue contractures).
  2. Children having visual or auditory defects.
  3. Children who can not understand verbal commands
  4. Children who had Botox application to the upper extremity in the past 6 months or had undergone a previous surgical intervention to wrist and hand.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
changes in upper limb functions | after 12 weeks of intervention
  using quality of upper extremity skills test (Quest)
changes in power grip strength | after 12 weeks of intervention
  using sphygmomanometer
changes in range of motion (ROM) | after 12 weeks of intervention
  using kinovea software

SECONDARY OUTCOMES:
changes in activity of daily living (ADL) | after 12 weeks of intervention
  using functional independence measure for children (WeeFIM):

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed B Ibrahim, Ass.Prof., Study Chair — head of pediatric department in faculty of physical therapy Kafrelshiekh university; Osama A El-Agamy, Professor, Study Director — Professor and head of department of pediatric department Faculty of medicine Kafrelshiekh university; Sara Y Abdel Elglil, Lecturer, Study Director — Lecturer in pediatric department in faculty of physical therapy Kafrelshiekh University
Locations (1):
- faculty of physical therapy Kafrelshiekh university, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atasavun Uysal S, Baltaci G. Effects of Nintendo Wii Training on Occupational Performance, Balance, and Daily Living Activities in Children with Spastic Hemiplegic Cerebral Palsy: A Single-Blind and Randomized Trial. Games Health J. 2016 Oct;5(5):311-317. doi: 10.1089/g4h.2015.0102. Epub 2016 Oct 5. PMID 27705006